CLINICAL TRIAL: NCT04724382
Title: Culturally-tailored Healthy Eating Education Intervention for Latinos in Massachusetts
Brief Title: Healthy Eating Education for Latinos
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Responsible Party: Principal Investigator, Josiemer Mattei, Donald and Sue Pritzker Associate Professor of Nutrition, Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IRB13-1332
Record Dates: First submitted 2021-01-22; First posted 2021-01-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Diet, Healthy; Diet Habit; Obesity; Blood Pressure; Psychological
MeSH Terms: conditions — Feeding Behavior; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants will be unaware of the which educational messages are considered intervention or control. Investigators will not be in contact with participants and will only receive coded data. Outcome assessor will be unaware of treatment allocation of participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Intervention group consisting of culturally-tailored healthy eating advice through daily text messages for 2 months (delivery phase). A reinforcement phase of 2-months will follow to repeat the text messages.
  Interventions: Behavioral: Culturally tailored healthy eating advice
- Control (Active Comparator): Control group consisting of general healthy eating advice through daily text messages for 2 months (delivery phase). A reinforcement phase of 2-months will follow to repeat the text messages.
  Interventions: Behavioral: Standard healthy eating advice

INTERVENTIONS:
Behavioral: Culturally tailored healthy eating advice — Culturally-tailored education includes strategies for healthy eating, preferences for traditional healthy foods, recommendations for limiting unhealthy traditional foods, portion sizes, etc.
  Arms: Intervention
Behavioral: Standard healthy eating advice — Standard healthy eating education includes strategies, foods, portions, and cooking and eating tips for general dietary recommendations
  Arms: Control

SUMMARY:
This intervention aims to evaluate the efficacy of a pilot educational intervention with deep-structure cultural tailoring for Latino ethnic groups on diet quality compared to general, surface-level healthy-eating messages.

ELIGIBILITY:
Inclusion Criteria:

* Aged 25-65 y/o
* Self-reported Hispanic/Latino heritage
* Able to understand and answer questions in Spanish or English
* Living in the Boston, MA metro area for the past 6 months and not planning to move in the next 6 months
* Has a cellphone with the capacity of receiving text messages and gives consent for the Study to text this number as part of the intervention

Exclusion Criteria:

* Younger than 25y or older than 65y
* Not Hispanic/Latino heritage
* Has condition or impairment that affects mental, cognitive, or memory abilities; such as Alzheimer's disease or stroke
* Has been diagnosed with cancer, diabetes (type 1 or 2), heart condition, major stomach condition (examples: coronary heart disease, heart attack, stroke or stroke, allergies, or severe diet restrictions)
* Does not understand Spanish or English
* Pregnant
* Under the care of an institution
* Living in another state outside of Massachusetts or planning to move in less than 6 months
* No cellphone with text capabilities (or cannot be used to receive texts from the Study)

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2019-04-29 (Actual); Primary Completion 2021-09-22 (Actual); Study Completion 2021-09-22 (Actual)

PRIMARY OUTCOMES:
Changes in diet quality score | 4 months
  Determine the change in score of short diet quality screener (range 18-54; from lowest to highest quality)
Changes in diet habits | 4 months
  Determine the change in the frequency of dietary behaviors (percent)

SECONDARY OUTCOMES:
Changes in diet satisfaction: diet satisfaction scale | 4 months
  Determine the change in the score of the Diet Satisfaction Questionnaire (DSat-45) (range 45-225; from lowest to highest satisfaction) and its summed seven subscales (ranges 5-40
Changes in attitude for eating: attitudes scale | 4 months
  Determine the change in the score of the attitudes scale (range 0-20; with positive and negative subscales for more attitudes towards healthy eating)
Changes in reasons for eating: reasons scale | 4 months
  Determine the change in the score of the reasons scale (range 0-15; fewer to more reasons to eat healthy)

OTHER OUTCOMES:
Changes in depression score: CESD | 4 months
  Determine the change in score of depressive symptom screener (range 0-54; from lowest to highest symptoms)
Change in levels of adipose risk factor | 4 months
  Estimate the change in the value of waist circumference (cm)
Change in levels of blood pressure risk factors | 4 months
  Estimate the change in the value of systolic and diastolic blood pressure (mmHg)
Changes in dysfunctional eating behaviors | 4 months
  Determine the change in score of the Three-Factor Eating Questionnaire (range 0-4; from lowest to highest dysfunctional eating and the three subscales of emotional, uncontrolled and restrictive eating behaviors)

CONTACTS AND LOCATIONS:
Locations (1):
- Harvard TH Chan School of Public Health, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD will be managed and distributed observing NIH and IRB policies on the dissemination and sharing of research results. Study information and requests for data will be available immediately upon the data being de-identified and properly revised for quality control by contacting study investigators.
Supporting Information: Study Protocol, ICF
Time Frame: 1 year
Access Criteria: The requested data will be shared with investigators via a secured, password-protected software website, upon request.

REFERENCES:
- [Derived] Mattei J, Caballero-Gonzalez A, Maafs-Rodriguez A, Zhang A, O'Neill HJ, Gago C. Lessons learned by adapting and implementing LUCHA: a deep-structure culturally tailored healthy eating randomized pilot intervention for ethnic-diverse Latinos. Front Public Health. 2024 Feb 20;11:1269390. doi: 10.3389/fpubh.2023.1269390. eCollection 2023. PMID 38445250